CLINICAL TRIAL: NCT01735604
Title: Pilot Study of Redirected Autologous T Cells Transduced to Express A CD20-Specific Chimeric Immunoreceptor in Patient With Chemotherapy Resistant or Refractory CD20+ Leukemia and Lymphoma
Brief Title: Genetically Engineered Lymphocyte Therapy in Treating Patients With Lymphoma That is Resistant or Refractory to Chemotherapy
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Han weidong, PI, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHN-PLAGH-BT-001
Record Dates: First submitted 2012-11-23; First posted 2012-11-28 (Estimated); Last update posted 2015-09-29 (Estimated); Status verified 2015-09

CONDITIONS: Hematopoietic/Lymphoid Cancer; Adult Acute Lymphoblastic Leukemia in Remission; B-cell Adult Acute Lymphoblastic Leukemia; B-cell Chronic Lymphocytic Leukemia; Prolymphocytic Leukemia; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Refractory Chronic Lymphocytic Leukemia; Stage III Adult Diffuse Large Cell Lymphoma; Stage III Chronic Lymphocytic Leukemia; Stage III Grade 1 Follicular Lymphoma; Stage III Grade 2 Follicular Lymphoma; Stage III Grade 3 Follicular Lymphoma; Stage III Mantle Cell Lymphoma; Stage IV Adult Diffuse Large Cell Lymphoma; Stage IV Chronic Lymphocytic Leukemia; Stage IV Grade 1 Follicular Lymphoma; Stage IV Grade 2 Follicular Lymphoma; Stage IV Grade 3 Follicular Lymphoma; Stage IV Mantle Cell Lymphoma
MeSH Terms: conditions — Hematologic Neoplasms; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Prolymphocytic; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Lymphoma, Mantle-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- anti-CD20-CAR T cell (Experimental): Arm 1 Patients receive anti-CD20-CAR lentiviral vector-transduced autologous T cells with 41BB vector for 3-5 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: anti-CD20-CAR vector-transduced autologous T cells; Other: genetically engineered lymphocyte therapy

INTERVENTIONS:
Biological: anti-CD20-CAR vector-transduced autologous T cells — anti-CD20-CAR vector-transduced autologous T cells
Other: genetically engineered lymphocyte therapy — genetically engineered lymphocyte therapy

SUMMARY:
RATIONALE: Placing a gene that has been created in the laboratory into white blood cells may make the body build an immune response to kill cancer cells.

PURPOSE: This clinical trial is studying genetically engineered lymphocyte therapy in treating patients with B-cell leukemia or lymphoma that is resistant or refractory to chemotherapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the safety and feasibility of the chimeric antigen receptor T cells transduced with the anti-CD20 vector (referred to as CART-20 cells).

II. Determine duration of in vivo survival of CART-20 cells. RT-PCR analysis of whole blood will be used to detect and quantify survival of CART-20 TCR zeta:4-1BB over time.

SECONDARY OBJECTIVES:

I. For patients with detectable disease, measure anti-tumor response due to CART-20 cell infusions.

II. Estimate relative trafficking of CART-20 cells to tumor in bone marrow and lymph nodes.

III. For patients with stored or accessible tumor cells (such as patients with active CLL, ALL, etc) determine tumor cell killing by CART-20 cells in vitro.

IV. Determine if cellular or humoral host immunity develops against the murine anti-CD20, and assess correlation with loss of detectable CART-20 (loss of engraftment).

V. Determine the relative subsets of CART-20 T cells (Tcm, Tem, and Treg).

OUTLINE: Patients are assigned groups according to order of enrollment.

Patients receive anti-CD20-CAR lentivirus vector-transduced autologous T cells with 41BB-gamma vector for 3-5 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed intensively for 6 months, every 3 months for 2 years, and annually thereafter for 13 years.

ELIGIBILITY:
Inclusion Criteria:

* •Male and female subjects with CD20+ B cell malignancies in patients with no available curative treatment options (such as autologous or allogeneic SCT) who have limited prognosis (several months to < 2 year survival) with currently available therapies will be enrolled

  * CD20+ leukemia or lymphoma
  * ALL in CR2 or CR3 and not eligible for allogeneic SCT because of age, comorbid disease, or lack of available family member or unrelated donor
  * Follicular lymphoma, previously identified as CD20+:
  * At least 2 prior combination chemotherapy regimens (not including single agent monoclonal antibody (Rituxan) therapy
  * Stage III-IV disease
  * Less than 1 year between last chemotherapy and progression (i.e. most recent progression free interval < 1 year)
  * Disease responding or stable after most recent therapy (chemotherapy, MoAb, etc)
  * CLL:
  * At least 2 prior chemotherapy regimens (not including single agent monoclonal antibody (Rituxan) therapy. Patients with high risk disease manifested by deletion chromosome 17p will be eligible if they fail to achieve a CR to initial therapy or progress within 2 years of 1 prior
  * Less than 2 years between last chemotherapy and progression (i.e. most recent progression free interval < 2 years)
  * Not eligible or appropriate for conventional allogeneic SCT
  * Patients who achieve only a partial response to FCR as initial therapy will be eligible.
  * Mantle cell lymphoma:
  * Beyond 1st CR with relapsed or persistent disease and not eligible or appropriate for conventional allogeneic or autologous SCT
  * Disease responding or stable after most recent therapy (chemotherapy, MoAb, etc...)
  * Relapsed after prior autologous SCT
  * B-cell prolymphocytic leukemia (PLL) with relapsed or residual disease after at least 1 prior therapy and not eligible for allogeneic SCT
  * Diffuse large cell lymphoma, previously identified as CD20+:
  * Residual disease after primary therapy and not eligible for autologous SCT
  * Relapsed after prior autologous SCT
  * Beyond 1st CR with relapsed or persistent disease and not eligible or appropriate of conventional allogeneic or autologous SCT
  * Expected survival > 12 weeks
  * Creatinine < 2.5 mg/dl
  * ALT/AST < 3x normal
  * Bilirubin < 2.0 mg/dl
  * Any relapse after prior autologous SCT will make patient eligible regardless of other prior therapy
  * Adequate venous access for apheresis, and no other contraindications for leukapheresis
  * Voluntary informed consent is given

Exclusion Criteria:

* •Pregnant or lactating women

  * The safety of this therapy on unborn children is not known
  * Female study participants of reproductive potential must have a negative serum or urine pregnancy test performed within 48 hours before infusion
  * Uncontrolled active infection
  * Active hepatitis B or hepatitis C infection
  * Concurrent use of systemic steroids. Recent or current use of inhaled steroids is not exclusionary
  * Previously treatment with any gene therapy products
  * Feasibility assessment during screening demonstrates < 30% transduction of target lymphocytes, or insufficient expansion (< 5-fold) in response to CD3/CD28 costimulation
  * Any uncontrolled active medical disorder that would preclude participation as outlined
  * HIV infection

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2013-01; Primary Completion 2017-05 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Occurrence of study related adverse events | Until week 24
  defined as >= Grade 3 signs/symptoms, laboratory toxicities, and clinical events) that are possibly, likely, or definitely related to study treatment

SECONDARY OUTCOMES:
Anti-tumor responses to CART-20 cell infusions | Baseline and post-infusion

CONTACTS AND LOCATIONS:
Locations (1):
- Biotherapeutic Department of Chinese PLA General Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Ernst M, Oeser A, Besiroglu B, Caro-Valenzuela J, Abd El Aziz M, Monsef I, Borchmann P, Estcourt LJ, Skoetz N, Goldkuhle M. Chimeric antigen receptor (CAR) T-cell therapy for people with relapsed or refractory diffuse large B-cell lymphoma. Cochrane Database Syst Rev. 2021 Sep 13;9(9):CD013365. doi: 10.1002/14651858.CD013365.pub2. PMID 34515338
- [Derived] Zhang WY, Wang Y, Guo YL, Dai HR, Yang QM, Zhang YJ, Zhang Y, Chen MX, Wang CM, Feng KC, Li SX, Liu Y, Shi FX, Luo C, Han WD. Treatment of CD20-directed Chimeric Antigen Receptor-modified T cells in patients with relapsed or refractory B-cell non-Hodgkin lymphoma: an early phase IIa trial report. Signal Transduct Target Ther. 2016 Mar 11;1:16002. doi: 10.1038/sigtrans.2016.2. eCollection 2016. PMID 29263894
- [Derived] Wang Y, Zhang WY, Han QW, Liu Y, Dai HR, Guo YL, Bo J, Fan H, Zhang Y, Zhang YJ, Chen MX, Feng KC, Wang QS, Fu XB, Han WD. Effective response and delayed toxicities of refractory advanced diffuse large B-cell lymphoma treated by CD20-directed chimeric antigen receptor-modified T cells. Clin Immunol. 2014 Dec;155(2):160-75. doi: 10.1016/j.clim.2014.10.002. Epub 2014 Oct 16. PMID 25444722